CLINICAL TRIAL: NCT05422183
Title: An Open, Single-arm Clinical Study of Envafolimab, Lenvatinib Combined With VP-16 in the Treatment of Platinum-resistant Recurrent Epithelial Ovarian Cancer，Primary Fallopian Tube Cancer and Primary Peritoneal Carcinoma
Brief Title: Envafolimab, Lenvatinib Combined With VP-16 in Platinum-resistant Recurrent Epithelial Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Yang Shen, chief physician, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENLEN-OC-001
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Ovarian Cancer, Epithelial
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — envafolimab; Immunotherapy; lenvatinib; Tyrosine Kinase Inhibitors; Etoposide; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- envafolimab，lenvatinib，VP-16 (Experimental): envafolimab：400mg，sc，d1，Q3W； lenvatinib：8 mg(BW<60 kg) OR 12 mg(BW≥60 kg)，po，qd，d1-21，Q3W； VP-16：50 mg/d, po,d1-14，Q3W
  Interventions: Drug: Envafolimab; Drug: Lenvatinib; Drug: VP-16

INTERVENTIONS:
Drug: Envafolimab — 400mg，sc，d1，Q3W
  Other Names: Immunotherapy
Drug: Lenvatinib — 8 mg(BW<60 kg) OR 12 mg(BW≥60 kg)，po，qd，d1-21，Q3W
  Other Names: Tyrosine kinase inhibitors
Drug: VP-16 — 50 mg/d, po,d1-14，Q3W
  Other Names: Chemotherapy

SUMMARY:
This study is a single-arm, open-label, exploratory clinical study, the main purpose is to evaluate the combination of envafolimab, lenvatinib VP-16 in the treatment of platinum-resistant recurrent epithelial ovarian cancer，primary fallopian tube cancer and primary peritoneal carcinoma.

DETAILED DESCRIPTION:
Platinum-resistant patients who have received at least 1 line chemotherapy in the past and the recurrence time is less than 6 months will receive envafolimab combined with lenvatinib and VP-16 for 6 cycles, followed by single-agent envafolimab maintenance therapy until disease progression, intolerable toxicity, or withdrawal of informed consent

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years；
* ECOG 0-1
* Life expectancy of at least 3 months；
* Histologically or pathologically confirmed epithelial ovarian cancer (EOC), fallopian tube cancer, primary peritoneal cancer； Ovarian cancer patients with drug-resistant recurrence after platinum-based chemotherapy；
* At least one measurable objective tumor lesion by spiral CT examination, the maximum diameter ≥ 1cm（according to RECIST 1.1）；
* Satisfactory main organ function，laboratory test must meet the following criteria: hemoglobin (HGB) ≥90g/L, neutrophil count（ANC） ≥1.5×109/L, platelet count（PLT） ≥80×109/L, Serum creatinine（CR）≤1.5 upper normal limitation (UNL)，total bilirubin (TBil) ≤1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 UNL (For patients with liver metastasis, the AST/ALT must be ≤5.0 UNL), Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN; left ventricular ejection fraction (LVEF) ≥ 50%; thyroid stimulating hormone (TSH) within the normal range Within: if the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
* Subjects of childbearing potential must use an appropriate method of contraception during the study period and within 120 days after the end of the study, have a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating subjects；

Exclusion Criteria:

* Suffered from other malignant tumors within 5 years before the start of treatment in this study;
* Grade ≥1 unresolved toxicities (according to the most recent version of the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE]) due to any prior therapy, excluding alopecia and fatigue; neurotoxicity was Recovery to ≤ grade 1 or baseline before the group;
* Subjects with any severe and/or uncontrolled disease ；
* Poorly controlled diabetes (fasting blood glucose [FBG] > 10 mmol/L) ；
* Received major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of study treatment; or had a long-term unhealed wound or fracture；
* Serious arterial/venous thrombotic event within 6 months prior to initiation of study treatment ；
* Previously received drug therapy against PD-1, PD-L1 and other related immune checkpoints ；
* Participating in or participating in other clinical investigators within 4 weeks prior to the start of the study ；
* Allergic to the active ingredients or excipients of the study drug ；
* Unsuitable for the study or other chemotherapy determined by investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  objective response rate

SECONDARY OUTCOMES:
OS | 12 months
  overall survival
PFS | 12 months
  progression free survival
DCR | 9 months
  disease control rate
AEs AEs | 12 months
  ａ advers adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yang Shen, MD, Study Director — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding B, Yu T, Zheng S, Xu J, Ji F, Lin H, Zhao X, Qiu S, Shen Y. Combination therapy for platinum-resistant ovarian cancer: a novel at-home regimen with envafolimab, lenvatinib, and etoposide. Oncologist. 2025 Sep 1;30(9):oyaf210. doi: 10.1093/oncolo/oyaf210. PMID 40658469